CLINICAL TRIAL: NCT04450043
Title: The Transitions Project: Supporting Adults During the Shift From Cancer Treatment to Surveillance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lara Traeger, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-140
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Non Small Cell Lung Cancer; Small-cell Lung Cancer; Mesothelioma; Cognitive Behavioral Therapy
Keywords: Non Small Cell Lung Cancer; Small-cell Lung Cancer; Mesothelioma; Cognitive Behavioral Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Mesothelioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Run In (Experimental): Participants will receive a 5-session psychoeducational intervention, focused on skills to enhance post-treatment quality of life with attention to (a) managing expectations, (b) coping with uncertainty, (c) self-managing residual symptoms and (d) strengthening social support.
  Interventions: Behavioral: Run-In Sessions 1-5
- Intervention (Experimental): Participants will receive a 5-session psychoeducational intervention, focused on skills to enhance post-treatment quality of life with attention to (a) managing expectations, (b) coping with uncertainty, (c) self-managing residual symptoms and (d) strengthening social support.
  Interventions: Behavioral: RCT Transitions Program Sessions 1-5
- Control (Active Comparator): Participants will receive a 1-session intervention, focused on reviewing goal progress for post-treatment quality of life, providing encouragement and support, identifying any current concerns, and providing tailored recommendations and resources.
  Interventions: Behavioral: RCT Control Session

INTERVENTIONS:
Behavioral: Run-In Sessions 1-5 — Session 1 explores patient goals and wishes for life after cancer treatment with a study interventionist. Sessions 2-5 focuses on learning and practicing skills to enhance post-treatment quality of life.
  Arms: Run In
Behavioral: RCT Transitions Program Sessions 1-5 — Sessions 1-5 focuses on learning and practicing skills to enhance post-treatment quality of life.
  Arms: Intervention
Behavioral: RCT Control Session — Participants will receive a 1-session intervention, focused on reviewing goal progress for post-treatment quality of life, providing encouragement and support, identifying any current concerns, and providing tailored recommendations and resources.
  Arms: Control

SUMMARY:
This research study is designed to develop and test a new supportive care program to help individuals with lung cancer improve their quality of life after cancer treatment is over.

DETAILED DESCRIPTION:
The aims of this pilot study are to evaluate the feasibility and acceptability of a brief psychoeducational intervention for participants with cancer who are transitioning from active treatment to surveillance.

The research study procedures include screening for eligibility.

This study consists of 2 parts. It is expected that about 45 people will take part in this research study.

* In the first part of this study, about 5 participants will complete survey questions and receive a 5-session program.
* In the second part of this study, about 40 participants will complete 3 surveys, and then will be randomly assigned to receive the 5-session program or to receive one study session (control).
* These sessions will focus on providing targeted support related to life after cancer treatment. The sessions will focus on skills for coping with uncertainty, managing symptoms, improving social support, and other topics important to the individual.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or older
* Diagnosis of non-small cell (NSCLC) or small cell (SCLC) lung cancer or mesothelioma
* Documented treatment plan with curative intent
* Ability to read and respond in English
* Treatment completion eligibility:

Run-in: Has completed treatment including systemic treatments and radiation as determined within the past three weeks by the cancer care team at Massachusetts General Hospital.

RCT: Has completed treatment including systemic treatments +/- radiation and +/- surgery.

1. If final treatment is systemic therapy +/- radiation: within three weeks after cancer care team determination that treatment is complete.
2. If final treatment is surgery: within three weeks after hospital discharge following surgery.

Exclusion Criteria:

* Comorbid health condition that would interfere with study participation
* Current participation in cognitive behavioral therapy treatment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants enrolled | 12 Weeks
  Feasibility will be assessed by calculating the proportions of potential participants enrolled (≥35%)
Number of participants retained | 12 Weeks
  Feasibility will be assessed by calculating the proportions of potential participants retained (≥70%)
Proportion of intervention arm participants who complete study visits | 12 weeks
  Feasibility will be assessed by calculating the proportion of intervention arm participants who complete study visits (≥70% attending ≥60% of sessions)

SECONDARY OUTCOMES:
Acceptability of study | Week 12
  Participant concerns and recommendations will be used to guide the next trial with respect to intervention content and delivery. Participant responses to the exit interview will be summarized (descriptive statistics for quantitative items) and coded (content analysis for open-ended items)
Change in Functional Assessment of Cancer Therapy-Lung Cancer (FACT-L) score | pre-baseline to 12 weeks
  This measure assesses multidimensional quality of life including physical well-being, social/family well-being, emotional well-being, functional well-being, and lung cancer-specific concerns. Each item is answered on a scale of 0 (not at all) to 5 (very much). Total scores will be used, with higher scores indicating better quality of life.
Change in Fear of Cancer Recurrence Scale 7 score | pre-baseline to 12 weeks
  This measure assesses worry about the return of disease with 6 items measured on a 5-point scale and 1 item measured on a 10-point scale. Total scores will be used, with higher scores indicating greater fear of recurrence.
Change in Hospital Anxiety and Depression Scale score | pre-baseline to 12 weeks
  This measure assesses depression and anxiety symptoms (7 items each), and mixed affect (all 14 items). Total scores will be used, with higher scores indicating greater distress.
Change in Multidimensional Scale of Perceived Social Support score | pre-baseline to 12 Weeks
  This measure assesses social support using 12 items on a 7-point Likert-type scale. Mean scores will be used, with higher scores indicating greater perceived support.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Traeger, Ph.D, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation